CLINICAL TRIAL: NCT01815814
Title: Therapeutic Potential of Myofascial Structural Integration in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Heidi M. Feldman, Ballinger-Swindells Professor of Developmental and Behavioral Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104644; 16807 (Other: Stanford University)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-05

CONDITIONS: Spastic Cerebral Palsy
Keywords: spasticity; cerebral palsy; hemiplegia; hemiparesis; diplegia; paraplegia; quadriplegia; quadriparesis
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Hemiplegia; Paresis; Paraplegia; Quadriplegia | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rolfing After 3-Month Wait (Experimental): The children in this arm receive the therapy (rolfing / myofascial structural integration) 3 months after they start the study.
  Interventions: Other: Rolfing / Myofascial Structural Integration
- Rolfing After 6-Month Wait (Other): The children in this arm receive the therapy (rolfing / myofascial structural integration) 6 months after they start the study.
  Interventions: Other: Rolfing / Myofascial Structural Integration

INTERVENTIONS:
Other: Rolfing / Myofascial Structural Integration — Rolfing is similar to deep massage. It is also known as "myofascial structural integration."

SUMMARY:
The investigators hypothesize that children with spastic cerebral palsy will show greater improvements in gross motor function, associated developmental skills and growth after the 3 months of myofascial structural integration treatment, a form of deep massage, than they showed after a 3- or 6-month pre-treatment waiting period.

The investigators further hypothesize that children with spastic CP will maintain their gains in gross motor function for ≥ 3 months after completion of MSI treatment.

DETAILED DESCRIPTION:
* The investigators will talk to you by telephone to determine if your child is eligible for the study.
* The study lasts for a total of 12 months with the massage treatment period lasting 12 weeks.
* The study entails a total of 10 sessions of Myofascial Structural Integration therapy over the 12-week period. Each session will last one hour.
* The child will have an evaluation of motor functions and development on enrollment and at three-month intervals for a total of 5 evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 up to, but not including, 7 years of age
* Children having the diagnosis of spastic cerebral palsy
* Children who have spasticity in one or both upper or lower limbs
* Children who are classified as either Gross Motor Function Classification System (GMFCS) level 2, 3 or 4 or Manual Ability Classification System (MACS) level 2, 3, 4 or 5

Exclusion Criteria:

* Children with active seizure disorders
* Children taking more than one medication to control their seizures
* Children with severe health problems that could be exacerbated by the treatment (such as severe chronic lung disease)
* Children who have undergone surgical treatments or botulinum injections within 6 months of entering the study
* Children who have planned surgical interventions during the studies time course
* Children with sensory, cognitive or language deficits which would affect their ability to understand directions necessary for assessment.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure Score | at Enrollment and every 3 months thereafter for up to 12 months

SECONDARY OUTCOMES:
Change in GAITRite Mat Measures | at Enrollment and every 3 months thereafter for up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Feldman, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Hansen AB, Price KS, Loi EC, Buysse CA, Jaramillo TM, Pico EL, Feldman HM. Gait changes following myofascial structural integration (Rolfing) observed in 2 children with cerebral palsy. J Evid Based Complementary Altern Med. 2014 Oct;19(4):297-300. doi: 10.1177/2156587214540466. Epub 2014 Jul 2. PMID 24989994
- See also: Click here for more information about this study — http://dbpresearch.stanford.edu